CLINICAL TRIAL: NCT01417286
Title: Accelerated, Hypofractionated Post-Mastectomy Radiation Therapy in Women With Breast Cancer: A Phase II Trial
Brief Title: Accelerated Radiation Therapy After Surgery in Treating Patients With Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Rutgers Cancer Institute of New Jersey (Other)
Responsible Party: Principal Investigator, Bruce G Haffty, Professor and Chairman, Department of Radiation Oncology Radiation Oncology, Rutgers, The State University of New Jersey
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 041001; NCI-2011-01124 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P30CA072720 (NIH); 0220100204 (Other: Rutgers IRB)
Record Dates: First submitted 2011-08-02; First posted 2011-08-16 (Estimated); Results first posted 2023-04-20 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-03

CONDITIONS: Inflammatory Breast Cancer; Invasive Ductal Breast Carcinoma; Invasive Lobular Breast Carcinoma; Mucinous Ductal Breast Carcinoma; Papillary Ductal Breast Carcinoma; Stage II Breast Cancer; Stage IIIA Breast Cancer; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer; Tubular Ductal Breast Carcinoma
MeSH Terms: conditions — Inflammatory Breast Neoplasms; Carcinoma, Ductal, Breast; Carcinoma, Lobular; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Radiation Therapy (Experimental): Patients undergo hypofractionated accelerated radiation therapy over 11 weekdays (for 15 elapsed days) within 21-63 days after last surgery or last course of chemotherapy. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Radiation: External beam radiation therapy

INTERVENTIONS:
Radiation: External beam radiation therapy — Hypofractionated accelerated radiation therapy over 11 days
  Other Names: EBRT

SUMMARY:
This phase II trial studies how well giving accelerated radiation therapy (RT) after surgery works in treating patients with breast cancer. RT uses high energy x rays to kill tumor cells. Giving RT after surgery may kill any remaining tumor cells

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Freedom from local failure and freedom from regional failure.

SECONDARY OBJECTIVES:

I. Acute toxicity and late toxicity using previously published toxicity scales. II. To identify co-variates responsible for poor cosmetic outcome in women with reconstructed chest walls when treated with accelerated, hypofractionated radiotherapy.

III. To correlate toxicity, cosmesis, and local control with molecular markers.

OUTLINE:

Patients undergo hypofractionated accelerated RT over 11 weekdays (for 15 elapsed days) within 21-63 days after last surgery or last course of chemotherapy. Treatment continues in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 2-8 weeks, every 3-6 months for 3 years, every 6-12 months for 2 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Invasive ductal, medullary, papillary, colloid (mucinous), or tubular histologies; invasive lobular carcinomas are allowed
* American Joint Committee for Cancer (AJCC) Stage IIa - IIIc (pathologic stage T0N1-3, T1N1-3, T2N1-3, T3N0-3, T4N0-3, all M0 status) histologically confirmed invasive carcinoma of the breast treated with mastectomy and either sentinel node biopsy or axillary dissection; inflammatory carcinoma (T4d) is allowed
* Patients with locally advanced breast cancer on clinical exam and diagnostics ( > 3 cm and/or clinically node-positive) who have mastectomy after induction chemotherapy are allowed
* Multifocal/multicentric disease is allowed
* Negative inked histologic margins of mastectomy (no invasive cells at margin) or positive margin at pectoralis fascia or skin
* Tamoxifen, Arimidex or other hormonal therapy is allowed; it may begin any time relative to the radiation at the discretion of the treating physician
* Chemotherapy is allowed, if chemotherapy is indicated the chemotherapy can be delivered first, followed by radiation therapy beginning 21-63 days after the last cycle of chemotherapy or the radiation therapy can be delivered first and the chemotherapy can be delivered no earlier than 21 days post radiation therapy; neoadjuvant chemotherapy is allowed; radiation therapy will be delivered after mastectomy or after any adjuvant chemotherapy as described above
* Chest wall reconstruction is allowed
* The patient must be enrolled and have treatment planning between 14-63 days from date of last surgery or last cycle of chemotherapy, and radiation must start within 21-63 days of date of last surgery or last cycle of chemotherapy
* Signed study-specific informed consent form prior to study entry
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1

Exclusion Criteria:

* Patient with distant metastases (M1)
* Patients with ductal or lobular carcinoma in-situ alone (no invasive component) and patients with non-epithelial breast malignancies such as sarcoma or lymphoma
* Patient with T1N0 or T2N0 disease
* Prior radiation therapy to the chest
* Patients with collagen vascular diseases, specifically systemic lupus erythematosus, scleroderma, or dermatomyositis
* Patients with co-existing medical conditions with life expectancy < 2 years
* Patients with psychiatric (with the possible exception of incompetence as defined by New Jersey [NJ] law) or addictive disorders that would preclude obtaining informed consent
* Other malignancy, except non-melanomatous skin cancer, < 5 years prior to participation in this study; the disease-free interval from any prior carcinoma must be continuous
* Women who are pregnant or lactating due to potential exposure of the fetus to RT and unknown effects of RT to lactating females
* Women who are able to conceive and unwilling to practice an effective method of birth control; women of childbearing potential must have a negative urine or serum pregnancy test within 7 days prior to treatment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2010-12-21 (Actual); Primary Completion 2020-02-20 (Actual); Study Completion 2020-02-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Haffty, MD, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (2):
- United States (2):
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Huntsman Cancer Hospital, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients enrolled at the Rutgers Cancer Institute of New Jersey and at the Huntsman Cancer Institute at the University of Utah. After enrolling 69 patients with stage II-III breast cancer, 67 women were eligible for analysis.
Period: Overall Study
Arm/Group | Radiation Therapy
Started | 67
Completed | 67
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Radiation Therapy
Number analyzed (Participants) | 67
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 60
  >=65 years | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 57
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 67

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Local, Regional, and/or Distant Failure
Description: Assessed by physical examination and other relevant imaging per the discretion of the patients treating physicians. Confirmed by biopsy, and should be coded as either chest wall recurrence, axilla, supraclavicular, or internal mammary.
Time Frame: Up to 5 years after dose of last treatment, an average of 62 months
Measure: Count of Participants; unit: Participants
Arm/Group | Radiation Therapy
Number analyzed (Participants) | 67
Participants | 12

2. Secondary Outcome: Count of Participants With Grade Three or Higher Toxicities
Description: Adverse events will be monitored weekly during treatment, then two weeks after RT, then at week 8, then every 3-6 months for 3 years, then every 6-12 months out to 5 years.
Time Frame: weekly during treatment, then two weeks after RT, then at week 8, then every 3-6 months for 3 years, then every 6-12 months out to 5 years.
Measure: Number; unit: participants
Arm/Group | Radiation Therapy
Number analyzed (Participants) | 67
participants | 7

3. Secondary Outcome: Participants With Plans for Breast Reconstruction, Having Grade Three or Higher Reconstruction Complications
Time Frame: Up to five years after dose of last treatment, an average of 62 months
Measure: Count of Participants; unit: Participants
Arm/Group | Radiation Therapy
Number analyzed (Participants) | 43
Participants | 15

ADVERSE EVENTS:
Time Frame: Up to five years after dose of last treatment, an average of 62 months
Arm/Group | Radiation Therapy
All-Cause Mortality (participants affected / at risk) | 6/67
Serious Adverse Events (participants affected / at risk) | 1/67
Other Adverse Events (participants affected / at risk) | 67/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radiation Therapy (N=67)
Infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radiation Therapy (N=67)
Dermatology/Skin (Skin and subcutaneous tissue disorders) | 38 (56)
Constitutional Symptoms (General disorders) | 35 (61)
Pain (General disorders) | 31 (83)
Neurology (Nervous system disorders) | 16 (20)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-10-18): https://cdn.clinicaltrials.gov/large-docs/86/NCT01417286/Prot_SAP_001.pdf
  • Informed Consent Form (2014-01-10): https://cdn.clinicaltrials.gov/large-docs/86/NCT01417286/ICF_000.pdf